CLINICAL TRIAL: NCT01699165
Title: Efficacy and Safety of Nasal Filters on Seasonal Allergic Rhinitis in a Double-blinded Randomized Placebo-controlled Crossover Pilot Study
Brief Title: Efficacy and Safety of Nasal Filters on Seasonal Allergic Rhinitis (Hay Fever)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Spirare ApS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1202-2; CIV-12-06-007121 (Other: Danish Health and Medicines Authority); 1-10-72-371-12. (Other: The Regional Ethics Committee on Biomedical Research, Central Denmark Region)
Record Dates: First submitted 2012-08-16; First posted 2012-10-03 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: rhinitis; allergic; seasonal; double blind; doubleblind; randomized; randomised; placebo; crossover; clinical; nasal; filter; controlled; trial; hayfever; hay; fever; efficacy; safety; prevention; adult; grass; pollen; symptom; Total nasal symptom score; acoustic rhinometry
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Nasal filter (Sham Comparator): Placebo treatment
  Interventions: Device: Placebo nasal filter
- Nasal Filter (Active Comparator): Active treatment
  Interventions: Device: Nasal filter

INTERVENTIONS:
Device: Nasal filter — Active nasal filter
  Arms: Nasal Filter
Device: Placebo nasal filter — Placebo nasal filter
  Arms: Placebo Nasal filter

SUMMARY:
The purpose of this study is to assess the effect of reducing exposure to allergens in patients with hay fever by means of a nasal filter.

ELIGIBILITY:
Inclusion Criteria:

* History of seasonal allergic rhinitis (SAR) for a minimum of 2 years before study entry. Documented by a positive skin test within 12 months of study enrollment.
* Written informed consent
* Reliable anticonception for fertile women
* Must be able to complete the study
* Forced Expiratory Volume at one second (FEV1) higher than 70 % of predicted value
* Positive grass immunoglobulin-E (IgE) blood sample equal to or higher than 3,50 kU/L

Exclusion Criteria:

* Positive pregnancy test for fertile women
* Asthma unless mild and only occurring in relation to the grass pollen season as assessed by the investigator
* Inadequate washout periods in regards to Environmental Exposure Unit (EEU) appointments (intranasal or systemic corticosteroids (1month), intranasal cromolyn (2 weeks), intranasal or systemic decongestants (3 days), intranasal or systemic antihistamines (3 days), loratadine (10 days))
* Rhinitis medicamentosa
* Use of long acting anti-histamines
* Documented evidence of acute or chronic sinusitis as determined by individual investigator
* FEV1 lower than 70 % of predicted value
* Subjects with perennial allergic rhinitis (PAR) to e.g. house dust mites, cats, dogs moulds unless symptom free
* Allergic rhinitis requiring medication caused by allergens other than grass unless symptom free
* Subjects with nasal conditions likely to affect the outcome of the study in the opinion of the investigator, i.e. anterior nasal septum deviation, nasal septum perforations, nasal polyps, chronic nasal obstruction or other nasal diseases
* Receipt of immunotherapy with grass pollen within the previous 10 years
* Women who are breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Effect of active nasal filters compared to placebo filters in the same patient group as measured by difference in maximum Total Nasal Symptom Score | Day 1 and day 15
  To assess the effects of active nasal filters on symptoms development in patients with seasonal allergic rhinitis (SAR) exposed to air-born allergens compared to the same patients in an exposed environment with a placebo nasal filter determined by their maximum Total Nasal Symptom Score (TNSS) out of the nine samples taken during a trial day. The statistical analysis will be done using non-parametric paired Wilcoxon signed rank test.

SECONDARY OUTCOMES:
Effect of active nasal filters compared to placebo filters as measured by acoustic rhinometry | Day 1 and day 15
  To assess the effects of active nasal filters on intranasal volume in patients with seasonal allergic rhinitis (SAR) exposed to air-born allergens compared to the same patients in an exposed environment with a placebo nasal filter. The assessment will be based on the difference between minimum and maximum volume as determined by acoustic rhinometry measurements pre- and post-exposure on each study day. The statistical analysis will be a parametric paired t-test.

OTHER OUTCOMES:
To assess symptoms using a VAS Scale symptoms questionnaire (PC) | Day 1 and Day 15
  On each study day: pre-exposure and post exposure: 30 minutes post and 3 hours post
To assess the tolerability and safety of nasal filters | Day 1 and Day 15
  By means of a product evaluation questionnaire. On each study day evaluated 30 minutes post exposure
To assess the effects on the lower airway via nitrogen oxide measurements during expiration. | Day 1 and Day 15
  On each study day: pre-exposure, 30 minutes post exposure and 3 hours post exposure
Spirometric lung function | Day 1 and Day 15
  On each study day: pre-exposure, 30 minute post exposure and in 3 hour intervals for 24 hours
Effect of active nasal filters compared to placebo filters in the same patient group as measured by difference in maximum Total Ocular Symptom Score (TOSS) | Day 1 and day 15
  To assess the effects of active nasal filters on symptoms development in patients with seasonal allergic rhinitis (SAR) exposed to air-born allergens compared to the same patients in an exposed environment with a placebo nasal filter determined by their maximum Total Ocular Symptom Score (TOSS) out of the nine samples taken during a trial day. The statistical analysis will be done using non-parametric paired Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Sigsgaard, Professor, Principal Investigator — Aarhus University, School of Public Health, Dept. of Environmental & Occupational Medicine
Locations (1):
- Aarhus University, School of Public Health, Department of Environmental & Occupational Medicine, Aarhus, Denmark